CLINICAL TRIAL: NCT04866654
Title: Radiation-Free Therapy for the Initial Treatment of Good Prognosis Early Non-bulky HL, Defined by a Low Metabolic Tumor Volume and a Negative Interim PET After 2 Chemotherapy Cycles- RAFTING
Brief Title: Radiation Free Chemotherapy for Early Hodgkin Lymphoma
Acronym: RAFTING
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBK132/1/2020
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Nivolumab, total dose 5760 mg milligram
  Interventions: Drug: Nivolumab 10 MG/ML

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — Nivolumab, 100 mg, 10 mg/ml

SUMMARY:
The results of the present study will provide information on short-term safety and efficacy of a iPET and MTV-adapted therapeutic strategy, aimed to assess the feasibility and safety on immediate disease control of a standard ABVD chemotherapy without any further treatment in patients with a very low risk or treatment failure. A second very important endpoint will be the efficacy of INRT "on demand" followed by Nivolumab maintenance for one year to rescue patients failing first-line treatment and relapsing with the pattern of "limited relapse" in terms of 3-Y failure from 2 relapse (FF2R). Patients entering into the study will be also asked to participate to a long-term follow up study (beyond ten years) to assess the prevalence of late-onset cardiovascular effects and secondary tumors in the cohort of patients enrolled in the experimental and control arm of the study. An exploratory endpoint has been also added such as the role of Minimal Residual Disease (MRD) detection by cell-free DNA assay on peripheral blood samples obtained during treatment in predicting long-term disease control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-60.
* Treatment-naïve, HL patients with Ann Arbor stage I or II A non-bulky disease stratified according to modified EORTC Criteria (refer to Appendix A);
* Patients must have histologically confirmed classical HL according to the current World Health Organization Classification (nodular sclerosis, mixed cellularity, lymphocytes rich, lymphocytes depleted, or classical HL NOS [not otherwise specified];
* ECOG performance status 0-2
* Hemoglobin must be > 8 gr./dL
* Absolute neutrophil count ≥ 1,000/μL
* Platelet count ≥ 100,000/μL
* Voluntary written consent to take part to the study
* Serum Creatinine < 2.0 mg/dL and/or Creatinine clearance or calculated Creatinine clearance > 40 mL/minute
* Total bilirubin must be < 2.0 x the upper limit of normal (ULN) unless known Gilbert syndrome
* ALT or AST must be < 3 x the upper limit of normal.
* Female patients: if postmenopausal for at least 1 year before enrolment or, if fertile - agreeing to practice 2 effective methods of contraception or agreeing to practice true abstinence.
* Male patients should agree to practice barrier contraception or to practice abstinence

Exclusion Criteria:

* Composite lymphoma or nodular lymphocyte-predominant Hodgkin lymphoma;
* Bulky disease (Lugano 2014 definition: single or conglomerated nodal mass with the largest diameter measuring 10 or more centimeters);
* B symptoms;
* Extra nodal site involved by disease;
* Female patients who are both lactating and breastfeeding or who have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug;
* Uncompensated diabetes mellitus requiring insulin therapy;
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol;
* Known human immunodeficiency virus (HIV) infection with a positive search for HIV antigens by immunoblot and/or circulating copies of HIV-RNA;
* Active hepatitis B with circulating copies of HBV-DNA, or active hepatitis C infection with circulating copies of HCV-RNA;
* Severely impaired, lung and renal function;
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection;
* Active autoimmune disorder in treatment with immunosuppressive drugs
* A left-ventricular ejection fraction < 50%;
* Myocardial infarction within 2 years of study entry.
* Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy exploration in terms of 3-Y PFS of chemotherapy alone | During follow-up (36 months) after the end of treatment
  To explore the efficacy, in terms of 3-Y PFS of chemotherapy alone in low-risk early-stage I-IIA HL patients, defined by both a low MTV and a negative interim PET after 2 courses of ABVD

SECONDARY OUTCOMES:
Efficacy exploration in terms of 3-Y PFS of chemotherapy plus Nivolumab | During follow-up (36 months) after the end of treatment
  To explore the efficacy in terms of 3-Y PFS of CMT plus Nivolumab in high-risk early-stage (I-IIA) HL (eHL), defined either by a positive PET- 2 or a high baseline MTV or both
Efficacy exploration in terms of 3-Y freedom from 2nd treatment failure (3-Y FF2TF) of chemotherapy followed by radiotherapy "on demand" plus Nivolumab maintenance | During follow-up (36 months) after the end of treatment
  To explore the efficacy in terms of 3-Y freedom from 2nd treatment failure (3-Y FF2TF) of chemotherapy followed by radiotherapy "on demand" plus Nivolumab maintenance in patients relapsing with the pattern of "limited relapse" (see below) for the entire group (relapsed and non-relapsed) of low-risk patients (with low MTV and negative PET- 2) high-risk early-stage (I-IIA) HL (eHL), defined either by a positive PET- 2 or a high baseline MTV or both
Safety exploration in terms of 3-Y OS of a treatment with chemotherapy alone | During follow-up (36 months) after the end of treatment
  To explore the safety in terms of 3-Y OS of a treatment with chemotherapy alone in low-risk early-stage (I-IIA) HL patients, defined by a low Metabolic Tumor Volume negative interim PET after 2 ABVD courses
Evaluation the ability of cell-free DNA (cfDNA) assay | During follow-up (36 months) after the end of treatment
  To evaluate the ability of cell-free DNA (cfDNA) assay to detect an impending relapse during follow-up in low-risk patients treated with chemotherapy alone�k�

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Zaucha, Professor, PhD, MD, Principal Investigator — Medical University of Gdansk; Andrea Gallamini, Professor, PhD, MD, Principal Investigator — Research and Clinical Innovation Department of the Lacassagne Cancer Center
Locations (27):
- Italy (12):
  - Hematology Department IRCCS Policlinico San Matteo, Pavia, P.le Golgi 19
  - Ospedale Papa Giovanni XXIII, Bergamo, Piazza OMS, 1
  - Istituto Europeo di Oncologia, Milan, Via Giuseppe Ripamonti 435
  - Hematology Department Azienda Ospedaliera S. Croce e Carle, Cuneo, Via Michele Coppino, 26
  - Azienda Ospedaliera Universitaria Policlinico Federico II, Napoli, Via S.Pansini, 5
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari, Viale Orazio Flacco, 65
  - Policlinico Università Tor Vergata, Roma, Viale Oxford, 81
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti, Ancona
  - Azienda Ospedaliera G. Brotzu - Ospedale Businco, Cagliari
  - Divisione Universitaria di Onco-Ematologia, Monza
  - Azienda Ospedaliera di Padova Dipartimento di Medicina Interna, Padua
  - Ospedali Riuniti Villa Sofia, Palermo
- Poland (4):
  - Gdański Uniwersytet Medyczny Department of Hematology and Transplantology, Gdansk
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Hematologii i Transfuzjologii ul. Indiry Gandhi 14 02-776 Warszawa, Warsaw
  - Uniwersyteckie Centrum Kliniczne im. Jana Mikulicza- Radeckiego we Wrocławiu, Wroclaw
- Spain (11):
  - Hospital Universitario Central de Asturias, Oviedo, Av. Roma
  - Hospital Universitario 12 de Octubre, Madrid, Avda de Córdoba
  - Hospital Duran i Reynals. Institut Catala d'Oncologia, Barcelona, Avinguda de La Granvia de l'Hospitalet, 199-203
  - Hospital Germans Trias i Pujol-ICO Badalona, Carretera de Canyet, Barcelona
  - Hospital Universitario Vall d'Hebron, Passeig de La Vall d'Hebron, 119-129, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, C. de Villarroel, 170
  - Hospital General Universitario Gregorio Marañon, Madrid, Calle Del Dr. Esquerdo
  - Hospital Universitario Marques de Valdecilla, Av. de Valdecilla, 25, Cantabria
  - Hospital Universitario Ramón y Cajal, Madrid, Ctra. de Colmenar Viejo Km. 9,100
  - Hospital Universitario de Salamanca, Salamanca, P.º de San Vicente, 58
  - Hospital Universitario Virgen del Rocio, Av. Manuel Siurot, Sevilla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712